CLINICAL TRIAL: NCT02232516
Title: Phase II Study of Romidepsin Plus Lenalidomide for Patients With Previously Untreated PTCL
Brief Title: Romidepsin and Lenalidomide in Treating Patients With Previously Untreated Peripheral T-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Celgene (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 14H04; NCI-2014-01770 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RV-CL-PTCL-PI-003974; STU00097620; P30CA060553 (NIH)
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Peripheral T-cell Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IIA Mycosis Fungoides/Sezary Syndrome; Stage IIB Mycosis Fungoides/Sezary Syndrome; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IIIA Mycosis Fungoides/Sezary Syndrome; Stage IIIB Mycosis Fungoides/Sezary Syndrome; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — romidepsin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (romidepsin, lenalidomide) (Experimental): Patients receive romidepsin IV over 4 hours on days 1, 8, and 15 and lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin; Drug: lenalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this study is to evaluate how safe and effective the combination of the study drugs romidepsin and lenalidomide is for treating patients with peripheral t-cell lymphoma (PTCL) who have not been previously treated for this cancer. Currently, there is no standard treatment for patients with PTCL; the most common treatment used is a combination of drugs called CHOP, but this can be a difficult treatment to tolerate because of side effects, and is not particularly effective for most patients with PTCL. Romidepsin (Istodax®) is a type of drug called an HDAC inhibitor. It interacts with DNA (genetic material in cells) in ways that can stop tumors from growing. It is given as an infusion through the veins. Lenalidomide (Revlimid®) is a type of drug known as an immunomodulatory drug, or IMID for short. This drug affects how tumor cells grow and survive, including affecting blood vessel growth in tumors. It is given as an oral tablet (by mouth).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of the combination of romidepsin plus lenalidomide in patients with previously untreated peripheral T-cell lymphoma (PTCL).

SECONDARY OBJECTIVES:

I. Evaluate the safety of the combination of romidepsin and lenalidomide. II. Further evaluate efficacy of the combination of romidepsin and lenalidomide.

III. Evaluate the delay to cytotoxic chemotherapy.

TERTIARY OBJECTIVES:

I. Evaluate the use of Northwestern Medicine (NM) positron emission tomography (PET)/computed tomography (CT) vs CT imaging in PTCL.

II. Validate a new prognostic model for newly diagnosed PTCL. III. Investigate the tumor immunohistochemical profile to identify potential biomarkers associated with prognosis and treatment response.

OUTLINE:

Patients receive romidepsin intravenously (IV) over 4 hours on days 1, 8, and 15 and lenalidomide orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 1 year in the absence of disease progression, inter-current illness that prevents further administration of treatment, unacceptable toxicity, patient decides to withdraw from study treatment (or study as a whole), or general or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the treating investigator.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of PTCL (using the most recent edition of the World Health Organization [WHO] Classification of Tumors of Hematopoietic and Lymphoid Tissues as guidance) including:

  * Anaplastic large cell lymphoma, anaplastic large cell kinase (ALK)-negative
  * Angioimmunoblastic T-cell lymphoma
  * Enteropathy-type T-cell lymphoma
  * Extranodal natural killer (NK)/T-cell lymphoma, nasal type
  * Hepatosplenic gamma-delta T-cell lymphoma
  * Peripheral T-cell lymphoma, unspecified (not otherwise specified [NOS])
  * Transformed mycosis fungoides
  * Subcutaneous panniculitis-like T-cell lymphoma.
  * NOTE: Patients with adequate archived (well-preserved, formalin-fixed) biopsy tissue remaining will be required to submit a portion for exploratory studies; this is not optional if tissue is available; however, lack of adequate tissue for exploratory studies will not preclude patients from participating
* Patients must have bi-dimensionally measurable disease (>= 1 cm) by CT imaging

  * NOTE: Patients with marrow-only disease are eligible; response for these patients will be assessed by repeat bone marrow biopsy
* Patients must fit into one of the following categories:

  * Age >= 18 years to < 60 years with a cumulative illness rating scale (CIRS) score >= 6 OR deemed ineligible for cytotoxic chemotherapy by the treating investigator
  * >= 60 years
* Patients must have adequate organ and marrow function (documented within 14 days prior to registration) as outlined below:

  * Absolute neutrophil count (ANC) >= 750/mcl
  * Hemoglobin >= 8 g/dl
  * Platelets >= 50,000/mcl
  * Total bilirubin =< 2 x upper limit normal (ULN)
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum pyruvate glutamate transaminase [SPGT]) =< 3 x ULN
  * Creatinine =< 2 x ULN
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* All patients must agree to use effective contraception while on study, and all patients must agree to undergo counseling sessions every 28 days about pregnancy precautions and risks of fetal exposure

  * Females of childbearing potential (FCBP) must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide, during lenalidomide therapy, during dose interruptions, and for at least 28 days following discontinuation of lenalidomide therapy
  * Males receiving lenalidomide must agree to use a latex condom during any sexual contact with FCBPs even if they have undergone a successful vasectomy
  * NOTE: A FCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
  * FCBP should be referred to a qualified provider of contraceptive methods, if needed
* FCPB must have a negative urine or serum pregnancy test within 7 days prior to registration, and be willing to adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategies (REMS®) program

  * NOTE: Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must be free of any prior malignancies for >= 1 year

  * NOTE: The exception to this would be currently treated squamous cell and basal cell carcinoma of the skin, carcinoma in situ of the cervix, breast, or bladder, or surgically removed melanoma in situ of the skin (stage 0) with histologically confirmed free margins of excision
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration

Exclusion Criteria:

* Patients with a diagnosis of any of the following are not eligible:

  * Anaplastic large cell lymphoma, ALK-positive
  * Adult T-cell lymphoma/leukemia (ATLL)
  * Anaplastic large-cell lymphoma, primary cutaneous type
  * Precursor T-lymphoblastic lymphoma/leukemia
  * Mycosis fungoides/Sezary syndrome (except transformed Mycosis fungoides [MF])
  * NK-cell leukemia
  * T-cell granular lymphocytic leukemia
  * T-cell prolymphocytic leukemia
* Patients must not have received prior systemic therapy for PTCL (except for corticosteroids for 10 or fewer days at any dose, no washout period required as long as they discontinue prior to starting study therapy); NOTE: topical treatment may have been given for prior existence of cutaneous lymphoma that has since become systemic PTCL; however, these topical therapies should be stopped at time of registration
* Patients who received chemotherapy (including monoclonal antibodies) or radiotherapy, administered for any condition, within 4 weeks prior to registration are not eligible
* Patients who received prior exposure to any other histone deacetylase (HDAC) inhibitors or immunomodulatory (IMID) agents for any reason are not eligible
* Patients receiving ongoing treatment with any other investigational agents are not eligible
* Patients who have known central nervous system (CNS) involvement of lymphoma are not eligible
* Patients who have an uncontrolled intercurrent illness including, but not limited to, any of the following are not eligible:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a known human immunodeficiency (HIV) infection are not eligible
* Patients who are pregnant or actively nursing an infant are not eligible
* Patients with a QT interval > 500 msec (using the Bazett's formula) within 28 days prior to registration are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2024-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Moreira, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Weill Cornell Medicine, New York, New York
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Ruan J, Zain J, Palmer B, Jovanovic B, Mi X, Swaroop A, Winter JN, Gordon LI, Karmali R, Moreira J, Petrich AM, Pro B. Multicenter phase 2 study of romidepsin plus lenalidomide for previously untreated peripheral T-cell lymphoma. Blood Adv. 2023 Oct 10;7(19):5771-5779. doi: 10.1182/bloodadvances.2023009767. PMID 37327113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population for this phase II study is patients with histologically confirmed (previously untreated) peripheral T-cell lymphoma (PTCL). Northwestern University will serve was the lead site and coordinating center for this study. Participating sites included Weill Cornell Medical College, and City of Hope. Enrollment began on 06/11/2015 at Northwestern University, 05/24/2017 at City of Hope, 12/14/2016 at Cornell University.
Period: Study Treatment Period: Cycles 1-3
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Started | 30
Cycle 1 | 29
Cycle 2 | 23
Cycle 3 | 20
1st Response Assessment | 23
Completed | 20
Not Completed | 10
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 1
Not completed — No Response | 1
Not completed — Screen failure | 1
Not completed — Disease Progression | 1
Period: Study Treatment Period: Cycles 4-6
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Started | 20
Cycle 4 | 15
Cycle 5 | 13
Cycle 6 | 13
2nd Response Assessment | 12
Completed | 13
Not Completed | 7
Not completed — Disease Progression | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Period: Study Treatment Period: Cycles 7-9
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Started | 13
Cycle 7 | 6
Cycle 8 | 4
Cycle 9 | 3
3rd Response Assessment | 3
Completed | 3
Not Completed | 10
Not completed — Adverse Event | 4
Not completed — Disease Progression | 2
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Period: Study Treatment Period: Cycles 10-12
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Started | 3
Cycle 10 | 3
Cycle 11 | 3
Cycle 12 | 1
Completed | 1
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1
Period: Survival Follow-up
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Started | 29
Completed | 5
Not Completed | 24
Not completed — Death | 15
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Still in follow-up | 5

BASELINE CHARACTERISTICS:
Population: One patient did not start any study treatment and was statistically withdrawn.
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 29
Age, Customized [Median (Full Range); unit: years]
  Age at Registration | 75 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 2
  Unknown or Not Reported | 3
Stage [Count of Participants; unit: Participants] — Ann Arbor Staging
  * I = Localized disease, single lymph node region or single organ
  * II = Two or more lymph node regions on the same side of diaphragm
  * III = Two or more lymph node regions above and below the diaphragm
  * IV = Widespread disease; multiple organs, with or without lymph node involvement
  Participants
    I | 1
    II | 1
    III | 14
    IV | 13
International Prognostic Index (IPI) Score [Median (Full Range); unit: units on a scale] — The International Prognostic Index (IPI) is a clinical tool developed by oncologists to aid in predicting the prognosis of patients with aggressive non-Hodgkin's lymphoma.
  One point is assigned for each of the following risk factors:
  * Age greater than 60 years
  * Stage III or IV disease
  * Elevated serum LDH
  * ECOG/Zubrod performance status of 2, 3, or 4
  * More than 1 extranodal site
  The sum of the points allotted correlates with the following risk groups:
  * Low risk (0-1 points)
  * Low-intermediate risk (2 points)
  * High-intermediate risk (3 points)
  * High risk (4-5 points)
  units on a scale | 3 [1 to 5]
Baseline LDH [Median (Full Range); unit: U/L] | 224 [110 to 868]
Subtype [Count of Participants; unit: Participants]
  Adult T-Cell Leukemia/lymphoma | 2
  Angioimmunoblastic T-cell Lymphoma | 16
  Enteropathy-type T-cell Lymphoma | 1
  Peripheral T-cell Lymphoma, unspecified | 10
International Prognostic Index (IPI) Score - Discrete [Count of Participants; unit: Participants] — The International Prognostic Index (IPI) is a clinical tool developed by oncologists to aid in predicting the prognosis of patients with aggressive non-Hodgkin's lymphoma.
  One point is assigned for each of the following risk factors:
  * Age greater than 60 years
  * Stage III or IV disease
  * Elevated serum LDH
  * ECOG/Zubrod performance status of 2, 3, or 4
  * More than 1 extranodal site
  The sum of the points allotted correlates with the following risk groups:
  * Low risk (0-1 points)
  * Low-intermediate risk (2 points)
  * High-intermediate risk (3 points)
  * High risk (4-5 points)
  Participants
    1 | 1
    2 | 6
    3 | 10
    4 | 11
    5 | 1
Bone Marrow Involvement [Count of Participants; unit: Participants]
  Indeterminate | 1
  Negative | 5
  Not Done | 16
  Positive | 7
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status
  * 0 = Fully active, able to carry on all pre-disease performance without restriction
  * 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work
  * 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  * 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  * 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  * 5 = Dead
  Participants
    0 | 8
    1 | 14
    2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), as Defined Per Cheson Criteria
Description: The endpoint for this objective will be objective response rate (ORR), defined per Cheson criteria. Response will be assessed by imaging after cycles 3 and 6, and then every 6 months thereafter. Response at 3 months (after cycle 3) will be used for purposes of the interim efficacy analysis.
Time Frame: Assessed after cycles 3 and 6, then every 6 months up to 3 years
Measure: Number; unit: participants
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 23
participants
  Complete Response (CR) | 6
  Partial Response (PR) | 9
  Stable Disease (SD) | 2
  Progressive Disease (PD) | 6
  CR + PR | 15

2. Secondary Outcome: Incidence of Toxicity Assessed Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The frequency and severity of toxicity events will be evaluated. All adverse events will be summarized as to type, severity, frequency, timing and attribution. Grade 3 or greater AEs that occurred in at least 10% of the patients are reported here
Time Frame: Evaluated once per cycle (1 cycle=28 days) up to 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 29
Participants
  Thrombocytopenia | 10
  Anemia | 8
  Lung Infection | 3
  Sepsis | 3
  Hypoalbuminemia | 7
  Fatigue | 5
  Hyponatremia | 13
  Hypertension | 11
  Hypokalemia | 4
  Hyperglycemia | 4
  Blood Bilirubin Increased | 4
  Dehydration | 3

3. Secondary Outcome: Progression-free Survival (PFS)
Description: l be progression-free survival (PFS)
  1 and 3 years after start of treatment as well as the duration of response from start of therapy, defined per Cheson criteria.
Time Frame: Reported at 1 and 3 years after the start of treatment
Measure: Number (95% Confidence Interval); unit: PFS Probability
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 23
PFS Probability
  PFS at year 1 | 0.486 [0.311 to 0.759]
  PFS at year 3 | 0.315 [0.108 to 0.615]

4. Secondary Outcome: Overall Survival (OS)
Description: Survival is defined as the duration of time from start of treatment to time of death, up to three years from the start of study treatment. Overall Survival (OS) is reported below as the proportion of patients who are alive at 1 and 2 years after starting treatment.
Time Frame: Reported at 1 and 2 years after the start of treatment
Measure: Number (95% Confidence Interval); unit: OS Probablilty
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 23
OS Probablilty
  OS at year 1 | 0.711 [0.540 to 0.937]
  OS at year 2 | 0.495 [0.316 to 0.778]

5. Secondary Outcome: Duration of Response, Defined Per Cheson Criteria
Description: The duration of overall response is measured from the time measurement criteria are met for Complete Remission or Partial Response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Assessed from start of therapy for up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 15
Days | 324 [8 to 1035]

6. Secondary Outcome: Delay to Cytotoxic Chemotherapy
Description: Time to first cytotoxic chemotherapy is defined as the time (in months) from start of study treatment to time of first dose of anti-neoplastic cytotoxic chemotherapy that is administered to treat lymphoma.
Time Frame: Up to 1 year
Population: This endpoint was not analyzed. No data was collected to analyze this endpoint.
Arm/Group | Treatment (Romidepsin, Lenalidomide)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: NM PET/CT vs. CT Imaging in PTCL
Description: To evaluate the use of NM PET/CT vs CT imaging in PTCL, a review of the utilized imaging modalities during treatment as a tool of response assessment will be done. When both imaging modalities are chosen for a patient, response assessment will be compared.
Time Frame: Up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Validate a New Prognostic Model for Newly Diagnosed PTCL
Description: Clinical biomarkers including age, race, histology, and stage as an assessment of prognosis. A points based system will be used to correlate with recently developed prognostic model.
Time Frame: Up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Immunohistochemistry Profile
Description: To investigate the tumor immunohistochemical profile to identify potential biomarkers associated with prognosis and treatment response. Archived tissue samples collected at baseline will be evaluated in order to determine how marker expression correlates with clinical outcome.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The reporting time frame for Adverse Events and Serious Adverse Events is from the time of consent through 30 days after treatment discontinuation, up to 1 year. The reporting time frame for All Cause Mortality is up to 2 years after staring treatment
Arm/Group | Treatment (Romidepsin, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 15/29
Serious Adverse Events (participants affected / at risk) | 23/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Romidepsin, Lenalidomide) (N=29)
Anemia (Blood and lymphatic system disorders) | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Death NOS (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 4
General disorders and administration site conditions - Other, specify (General disorders) | 3
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Lung infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Romidepsin, Lenalidomide) (N=29)
Anemia (Blood and lymphatic system disorders) | 26
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Lymph node pain (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 8
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 3
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Anal pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic hemorrhage (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 19
Diarrhea (Gastrointestinal disorders) | 14
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 22
Oral dysesthesia (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 7
Edema face (General disorders) | 2
Edema limbs (General disorders) | 12
Fatigue (General disorders) | 20
Fever (General disorders) | 11
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 5
Hypothermia (General disorders) | 1
Injection site reaction (General disorders) | 1
Localized edema (General disorders) | 4
Malaise (General disorders) | 1
Multi-organ failure (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 5
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 3
Immune system disorders - Other, specify (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 6
Fall (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 14
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 12
Electrocardiogram QT corrected interval prolonged (Investigations) | 3
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 6
Lymphocyte count decreased (Investigations) | 26
Neutrophil count decreased (Investigations) | 20
Platelet count decreased (Investigations) | 27
Weight loss (Investigations) | 13
White blood cell decreased (Investigations) | 20
Anorexia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 26
Hypocalcemia (Metabolism and nutrition disorders) | 22
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 18
Hypomagnesemia (Metabolism and nutrition disorders) | 19
Hyponatremia (Metabolism and nutrition disorders) | 26
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 11
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 8
Confusion (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 7
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 20
Hypotension (Vascular disorders) | 7
Lymphedema (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02232516/Prot_SAP_000.pdf